CLINICAL TRIAL: NCT03181113
Title: A Multi-center, Prospective Study to Acess Long-term Benefit in HBeAg Positive Chronic Hepatitis B Patients Who Previously Received Standard Peginterferon Alfa Therapy
Brief Title: Long-term Benefit in Chronic Hepatitis B Patients After Standard Peginterferon Alfa Therapy
Status: Completed | Type: Observational
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TB1510IFN
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B
Keywords: peginterferon alpha; HBeAg seroconversion; immune control
MeSH Terms: conditions — Hepatitis B | interventions — peginterferon alfa-2b; peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, hemocyte
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- peginterferon alfa 2b
  Interventions: Drug: Peginterferon Alfa-2B
- peginterferon alfa 2a
  Interventions: Drug: Peginterferon Alfa-2A

INTERVENTIONS:
Drug: Peginterferon Alfa-2B — pre-received standard peginterferon alfa-2b therapy
  Other Names: pegberon
  Groups: peginterferon alfa 2b
Drug: Peginterferon Alfa-2A — pre-received standard peginterferon alfa-2a therapy
  Other Names: pegasys
  Groups: peginterferon alfa 2a

SUMMARY:
In this cohort study, patients with chronic hepatitis B who prior participated in TB1211IFN study and received at least 39 doses of peginterferon alfa will be enrolled. HBsAg/anti-HBs level, HBeAg/anti-HBe level, Serum HBV DNA load and alanine transaminase level will be test every year from the second year to the fifth year after the ending of peginterferon alfa treatment, and long-term benefit of interferon treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign the informed consent form.
* Participated in NCT01760122 study (TB1211IFN) and has received at least 39 doses of peginterferon.

Exclusion Criteria:

* Conditions which in the opinion of the investigator should be precluded from the study(e.g., poor compliance).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B who previously participated in TB1211IFN study.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
rate of HBeAg seroconversion | from the second year to the fifth year

SECONDARY OUTCOMES:
decent degree of HBeAg | from the second year to the fifth year
decent degree of HBV DNA | from the second year to the fifth year
rate of alanine aminotransferase normalization | from the second year to the fifth year
rate of HBeAg loss | from the second year to the fifth year
rate of HBV DNA undetectable | from the second year to the fifth year
rate of HBeAg seroconversion | from the second year to the fifth year

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, MD, Principal Investigator — Peking University First Hospital
Locations (28):
- China (28):
  - 302 Military Hospital, Beijing, Beijing Municipality
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital Chongqing Medical University, Chongqing, Chongqing Municipality
  - Southwest Hospital, Chongqing, Chongqing Municipality
  - Fuzhou Infectious Disease Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Xiamen Hospital of T.C.M, Xiamen, Fujian
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Beijing University Shenzhen Hospital, Shenzhen, Guangdong
  - Third Affiliated Hospital, Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital, Central-south University, Changsha, Hunan
  - Xiangya Second Hospital, Central-south University, Changsha, Hunan
  - 81 Military Hospital, Nanjing, Jiangsu
  - Second Hospital of Nanjing, Nanjing, Jiangsu
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shenyang Sixth People's Hospital, Shenyang, Liaoning
  - Jinan Infectious Disease Hospital, Jinan, Shandong
  - 85 Military Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Ruijing Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Tianjin Third Central Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No